CLINICAL TRIAL: NCT00001022
Title: A Randomized, Comparative Trial of Zidovudine (AZT) Versus AZT Plus Didanosine (ddI) Versus AZT Plus Dideoxycytidine (ddC) in HIV-Infected Patients
Brief Title: A Comparison of Zidovudine (AZT) Used Alone or in Combination With Didanosine (ddI) or Dideoxycytidine (ddC) in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: CPCRA 007; 11559 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; Zalcitabine; Didanosine

INTERVENTIONS:
Drug: Zidovudine
Drug: Zalcitabine
Drug: Didanosine

SUMMARY:
Primary: To compare the efficacy of zidovudine ( AZT ) given alone versus AZT plus didanosine ( ddI ) versus AZT plus zalcitabine ( dideoxycytidine; ddC ) in delaying the occurrence of AIDS-related conditions in HIV-infected patients.

Secondary: To compare the frequency and severity of adverse experiences in the three regimens. To compare the mortality rates in the three regimens. To compare the effects of antiretroviral regimens on CD4+ cell levels.

Studies have indicated that maintenance therapy with AZT over extended periods may be limited by dose-dependent toxicity, primarily myelosuppression, and by the emergence of drug-resistant HIV strains. It is anticipated that the combination of AZT with either ddI or ddC may promote higher antiviral efficacy, with acceptable toxicity and less likelihood of development of drug-resistant strains, than AZT alone.

DETAILED DESCRIPTION:
Studies have indicated that maintenance therapy with AZT over extended periods may be limited by dose-dependent toxicity, primarily myelosuppression, and by the emergence of drug-resistant HIV strains. It is anticipated that the combination of AZT with either ddI or ddC may promote higher antiviral efficacy, with acceptable toxicity and less likelihood of development of drug-resistant strains, than AZT alone.

Approximately 1200 patients are randomized in a 2:1:1:2 ratio to one of the following four treatment arms: AZT plus ddI, AZT plus ddI placebo, AZT plus ddC placebo, and AZT plus ddC. Average follow-up is 2 years.

ELIGIBILITY:
Inclusion Criteria

Required:

* Documented HIV infection OR working diagnosis of HIV OR evidence of idiopathic suppression with an AIDS-defining opportunistic infection or malignancy (except Kaposi's sarcoma).
* CD4+ cell count = or < 200/mm3 or = or < 15 percent of total lymphocyte count within previous 90 days OR history of AIDS-defining opportunistic infection.
* Current PCP prophylaxis.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Symptoms of pancreatitis or peripheral neuropathy of grade 2 or worse.
* Requirement for acute therapy for any active AIDS-defining opportunistic infection or systemic chemotherapy for malignancy.
* Stage 2 or worse (moderate) AIDS Dementia Complex.
* Other disorders or conditions for which the study drugs are contraindicated or that may prevent adequate compliance with study therapy.

Concurrent Medication:

Excluded:

* Acute therapy for active AIDS-defining opportunistic infection.
* Systemic chemotherapy for malignancy.
* Antiretroviral therapy other than that provided by this study.

Patients with the following prior conditions are excluded:

* History of pancreatitis or peripheral neuropathy of grade 2 or worse.
* History of intolerance to the study drugs at entry doses and/or frequencies.
* History of phenylketonuria.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200
Dates: Study Completion 1995-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L Saravolatz, Study Chair; D Winslow, Study Chair
Locations (16):
- United States (16):
  - Community Consortium of San Francisco, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Hill Health Corp, New Haven, Connecticut
  - Wilmington Hosp / Med Ctr of Delaware, Wilmington, Delaware
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Addiction Research and Treatment Corp, Brooklyn, New York
  - Clinical Directors Network of Region II, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Richmond AIDS Consortium, Richmond, Virginia

REFERENCES:
- [Background] New trials reach same conclusion: two drugs are better than AZT alone. AIDS Alert. 1995 Nov;10(11):133-6. PMID 11362921
- [Background] Saravolatz LD, Collins G, Hodges D, Winslow D, Pettinelli C. A randomized, comparative trial of ZDV versus ZDV plus ddI versus ZDV plus ddC in persons with CD4 cell counts of less than 200/mm3. Int Conf AIDS. 1996 Jul 7-12;11(1):21 (abstract no MoB291)
- [Background] Ethnicity and treatment. Proj Inf Perspect. 1997 Jul;(22):15-6. PMID 11364573
- [Background] Besch CL, Morse E, Simon P, Hodges J, Franchino B. Preliminary results of a compliance study within CPCRA 007 combination nucleoside study (NuCombo). Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:111 (abstract no 254)
- [Background] Mayers D, Saravolatz L, Winslow D, Jagodzinski L, Collins G, Hodges D, Pettinelli C, Weislow O, Stein D. Viral burden measurements in CPCRA 007. Int Conf AIDS. 1996 Jul 7-12;11(Program Supplement):16 (abstract no ThB911)
- [Background] Kumi J, Collins G, Saravolatz L. Does ethnicity influence the efficacy and toxicity of combination versus monotherapy with nucleosides in AIDS patients? Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:166 (abstract no 547)
- [Background] James JS. AZT, ddI, and ddC combinations at FDA advisory hearing. Food and Drug Administration. AIDS Treat News. 1996 Apr 5;(no 244):6. PMID 11363307
- [Background] Researchers are rethinking role of AZT in drug therapy. AIDS Policy Law. 1995 Oct 6;10(18):11. PMID 11362821
- [Background] Saravolatz LD, Winslow DL, Collins G, Hodges JS, Pettinelli C, Stein DS, Markowitz N, Reves R, Loveless MO, Crane L, Thompson M, Abrams D. Zidovudine alone or in combination with didanosine or zalcitabine in HIV-infected patients with the acquired immunodeficiency syndrome or fewer than 200 CD4 cells per cubic millimeter. Investigators for the Terry Beirn Community Programs for Clinical Research on AIDS. N Engl J Med. 1996 Oct 10;335(15):1099-106. doi: 10.1056/NEJM199610103351503. PMID 8813040
- [Background] Randall P. CPCRA 007: preliminary results of combination antiretroviral study. NIAID AIDS Agenda. 1996 Mar:2. PMID 11363796
- [Derived] Niu F, Zheng C, Liu L. Exploring causal mechanisms and quantifying direct and indirect effects using a joint modeling approach for recurrent and terminal events. Stat Med. 2023 Sep 30;42(22):4028-4042. doi: 10.1002/sim.9846. Epub 2023 Jul 17. PMID 37461207